CLINICAL TRIAL: NCT02009631
Title: A Randomized, Placebo-Controlled Crossover Study to Evaluate the Effect of Veliparib (ABT-888) on Cardiac Repolarization in Subjects With Relapsed or Refractory Solid Tumors
Brief Title: A Study to Evaluate the Effects of Veliparib on Heart Rhythms in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: M12-020; 2013-002028-18 (EudraCT Number)
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2014-12

CONDITIONS: Breast Cancer; Ovarian Cancer; Colon Cancer; Lung Cancer; Gastric Cancer; Solid Tumors
Keywords: Solid Tumors; Ovarian Cancer; Colon Cancer; Lung Cancer; Breast Cancer; Gastric Cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Colonic Neoplasms; Lung Neoplasms; Stomach Neoplasms | interventions — veliparib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sequence Group A (Experimental): 200 mg Veliparib
  Interventions: Drug: Veliparib (ABT-888)
- Sequence Group B (Experimental): 400 mg Veliparib
  Interventions: Drug: Veliparib (ABT-888)
- Sequence Group C (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Veliparib (ABT-888)
  Arms: Sequence Group A; Sequence Group B
Drug: Placebo
  Arms: Sequence Group C

SUMMARY:
This is a randomized Phase 1 study to evaluate the effects of Veliparib on cardiac repolarization in patients with solid tumors who's cancer has recurred or is no longer responding to current treatment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed solid malignancy that is metastatic or unresectable for which standard curative measures or other therapy that may provide clinical benefit do not exist or are no longer effective.
* Subjects with brain metastases must have clinically controlled neurologic symptoms.
* Subject is able to swallow and retain oral medications and does not have uncontrolled emesis.
* Subject has adequate bone marrow, renal and hepatic function per local laboratory reference ranges.

Exclusion Criteria:

* Uncorrected serum potassium, serum magnesium, serum calcium or free thyroxin (FT4) and thyroid stimulating hormone (TSH) outside of normal reference ranges, or grade 2 hyponatremia or hypernatremia.
* Subject has severe ECG morphologic abnormalities that make QTc evaluation difficult.
* Subject has a history of cardiac conduction abnormalities.
* Subject has a significant history of cardiovascular disease.
* Subject has received any anti-cancer therapies 21 days prior to the first dose of study drug, or has recovered to no better than a grade 2 or higher clinically significant adverse effect(s)/toxicity(s) of the previous therapy.
* Use of drugs with a known risk for QT prolongation and Torsades de Pointes within 7 days prior to the first study dose.
* Use of tobacco or nicotine-containing products within 12 hours prior to the first study dose.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of Veliparib on corrected QT interval calculated by Fridericia's formula (QTcF) | Electrocardiograms (ECGs) will be done at Screening, 6 time points on Day 1 of Periods 1, 2 and 3 in triplicate, 1 time point on Day 2 of Periods 1, 2, and 3 and 1 time point on Day 3 of Period 3.

SECONDARY OUTCOMES:
Pharmacokinetic sampling maximum observed plasma concentration (Cmax) | Pharmacokinetic samples will be drawn at Screening, 6 time points on Day 1 of Periods 1, 2 and 3 and 1 time point on Day 2 of Periods 1, 2, and 3.
Pharmacokinetic sampling - time to maximum observed plasma concentration (Tmax) | Pharmacokinetic samples will be drawn at Screening, 6 time points on Day 1 of Periods 1, 2 and 3 and 1 time point on Day 2 of Periods 1, 2, and 3.
Pharmacokinetic sampling - the area under the plasma concentration-time curve (AUC) from time 0-24 hours (AUC 0-24) | Pharmacokinetic samples will be drawn at Screening, 6 time points on Day 1 of Periods 1, 2 and 3 and 1 time point on Day 2 of Periods 1, 2, and 3.
The number of subjects with adverse events | Up to 30 days after last dose of study drug.
Vital Signs | Up to 30 days after last dose of study drug.
  Blood pressure, heart rate and temperature.
Clinical Laboratory Tests | Up to 30 days after last dose of study drug.
  Hematology, chemistry, urinalysis
Tumor Assessment | Screening
  A computerized tomography scan will be done at screening to document tumor size.

CONTACTS AND LOCATIONS:
Overall Officials: Stacie Shepherd, PhD, Study Director — AbbVie
Locations (5):
- United States (2):
  - Site Reference ID/Investigator# 116015, Scottsdale, Arizona
  - Site Reference ID/Investigator# 116016, San Antonio, Texas
- Netherlands (2):
  - Site Reference ID/Investigator# 117320, Groningn
  - Site Reference ID/Investigator# 117336, Maastricht
- Site Reference ID/Investigator# 117517, Madrid, Spain

REFERENCES:
- [Result] Munasinghe W, Stodtmann S, Tolcher A, Calvo E, Gordon M, Jalving M, de Vos-Geelen J, Medina D, Bergau D, Nuthalapati S, Hoffman D, Shepherd S, Xiong H. Effect of veliparib (ABT-888) on cardiac repolarization in patients with advanced solid tumors: a randomized, placebo-controlled crossover study. Cancer Chemother Pharmacol. 2016 Nov;78(5):1003-1011. doi: 10.1007/s00280-016-3156-x. Epub 2016 Oct 5. PMID 27709282